CLINICAL TRIAL: NCT01632787
Title: Utility of a Survey Instrument to Predict Benefit From a Novel Treatment for Vertical Heterophoria
Acronym: VH
Status: Completed | Type: Observational
Sponsor: Vision Specialists of Birmingham (Other)
Collaborators: Trinity Health Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: VSofM 4-2012
Record Dates: First submitted 2012-05-15; First posted 2012-07-03 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Binocular Vision Dysfunction; Vertical Heterophoria
Keywords: Anxiety; Binocular; Chronic Headache; Dizziness; Vertical Heterophoria; Vision Dysfunction
MeSH Terms: conditions — Anxiety Disorders; Headache Disorders; Dizziness; Vision Disorders | interventions — Surveys and Questionnaires; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaires and Optometrist Prism Challenge/Treatment — A Vertical Heterophoria Symptom Questionnaire (VHSQ) as well as Headache Disability Index (HDI) survey is used on all Emergency Department (ED) headache patients to assess medical history and symptom burden. Prism testing (or Prism Challenge) is performed by the study optometrist to identify those who have Vertical Heterophoria (VH). Prism Challenge is similar to prescription eyeglass testing, but with unique lenses that are meant to reduce strain on eyes that are misaligned. Follow-up questionnaires are then administered to assess any improvement in symptom burden.

SUMMARY:
Patients with acute exacerbation of chronic headache disorder present frequently to the Emergency Department (ED) for pain management. A novel etiology of headaches is Vertical Heterophoria (VH), a poorly understood and little recognized binocular vision malady that when treated with realigning prismatic spectacle lenses results in marked reduction in headache and other associated VH symptoms.

This study aims to determine the accuracy of the Vertical Heterophoria Symptom Questionnaire (VHSQ) in identifying a ED headache patients who will experience significant reduction in VH symptoms with use of realigning prismatic spectacle lenses. This study's secondary purpose is to determine if VH is a common cause of chronic headache disorders in ED headache patients.

To achieve these goals, a prospective observational study will be performed on ED headache patients > 18 years old. All will be given the VHSQ, and all will be assessed for a diagnosis of VH by an optometrist who will utilize a novel VH testing method. High and low score groups on the VHSQ will then be compared to each other to determine the prevalence of VH in each.

ELIGIBILITY:
Initially include all patients presenting to Emergency Department with chief complaints of Headache, Head Pain, Face Pain and/or Migraine.

Inclusion Criteria:

* Greater than or equal to 18 years old
* Ability to speak and read English
* Chronic headache disorder as defined by physician diagnosis, or greater than three months of headaches requiring symptom relief with medication more than once every two weeks, or having headaches so severe that previous Emergency Department evaluation or treatment was necessary

Exclusion Criteria:

* Symptoms directly caused by trauma within the last three months
* Known TMJ disorder and presenting with TMJ pain
* Suspected infectious sinusitis or meningitis
* Pain originating from ear
* Pain originating from dental source
* Patient not willing or able to travel to study optometrist for follow-up
* Known history of cerebral aneurysm
* Known history of brain tumor
* Without previous CT, MRI, or other imaging to assess patient's headache disorder
* Patient a prisoner
* Patient under temporary or permanent custodianship
* Patient currently with questionable state of mental competence
* Treating physician or study investigator believes patient to be inappropriate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the Emergency Department at St. Joseph Mercy Hospital with complaint of non-traumatic exacerbation of chronic headaches of previously unknown etiology.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2012-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
VH Diagnosis | 2-4 Weeks
  Significant reduction of symptom burden as reflected on follow-up Severity Index (SI) score with prismatic spectacle challenge and treatment.
VH Diagnosis | 2-4 Weeks
  Significant reduction of symptom burden as reflected on follow-up Vertical Heterophoria Symptom Questionnaire (VHSQ) score with prismatic spectacle challenge and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Rosner, MD, Principal Investigator — St. Joseph Mercy Hospital; Debra Feinberg, OD, Study Director — Vision Specialists of Michigan
Locations (2):
- United States (2):
  - Vision Specialists of Michigan, Bloomfield Hills, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan

REFERENCES:
- See also: Related Info — http://www.VSofM.com